CLINICAL TRIAL: NCT03339843
Title: Multiorgan Metabolic Imaging Response Assessment of Abemaciclib
Acronym: MiMe-A
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jules Bordet Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IJB-MULTI-MIME-A-2017
Record Dates: First submitted 2017-10-05; First posted 2017-11-13 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-07

CONDITIONS: Esophageal Adenocarcinoma; Esophagus SCC; Cholangiocarcinoma; Urothelial/Bladder Cancer, Nos; Endometrial Cancer
Keywords: cancer
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Cholangiocarcinoma; Urologic Neoplasms; Endometrial Neoplasms; Neoplasms | interventions — abemaciclib

STUDY DESIGN:
Intervention Model Description: This is a two step, open-label, basket trial looking at 5 different tumour types.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abemaciclib (Experimental): This study contains 2 stages; during the 1st stage, a maximum of 17 patients will be enrolled in each tumour type cohort. After 13 evaluable patients have been enrolled, an interim analysis will be performed. If 3 or more patients are seen to have experienced a treatment success, then the cohort will pass into the 2nd stage in which a maximum of 20 more patients are enrolled. If 2 or less patients are seen to have experienced a treatment success, then that cohort will be closed and will not proceed into the 2nd stage.
  Subjects will receive 200 mg of abemaciclib orally, twice a day, during cycles of 28 days each. The subject will undergo: A baseline FDG-PET/CT and a baseline CT scan and A blinded early FDG-PET/CT at D14 +/- 2 days of study treatment.
  A treatment success is defined as a patient who has metabolic response according to PERCIST with a response cut off set at 15% at the early FDG-PET/CT and a morphological disease control after 2 cycles measured by RECIST v1.1.
  Interventions: Drug: Abemaciclib

INTERVENTIONS:
Drug: Abemaciclib — Subjects will receive 200 mg of abemaciclib orally, two times a day, during cycles of 28 days each. An early FDG-PET/CT will be performed at cycle 1 day 14 to search for any new lesions.
  Other Names: FDG-PET/CT

SUMMARY:
Open-label, phase II, basket trial. This trial is a screening program for abemaciclib efficacy in multiple platinum-resistant tumour types by using metabolic imaging (PERCIST) and RECIST v1.1 criteria.

Based on the rate of FDG-avidity and the absence of deactivation of the Rb gene function in more than 95% of cases, we propose to define 5 tumour types of interest in a preliminary stage:

1. Platinum-refractory esophageal adenocarcinoma (ADC)
2. Platinum-refractory esophageal squamous cell carcinoma (SCC)
3. Platinum-refractory cholangiocarcinoma
4. Platinum-refractory and progressive after immunotherapy urothelial cancer
5. Platinum-refractory endometrial cancer

DETAILED DESCRIPTION:
In various solid tumour types FDG-PET/CT has been shown to identify treatment-refractory diseases with a high negative predictive value (NPV) through a whole-body quantitative assessment of treatment-induced changes in tumour glucose uptake soon after treatment initiation, before any structural changes are observed. Progress in the standardisation of FDG-PET/CT imaging and response analysis now allow its use in multicentric trials opening the possibilities for trials where treatment allocation will be based on early metabolic response. MiMe has been built on the assumption that a medication which does not induce any metabolic changes in a given clinical setting is unlikely to induce a significant benefit and does consequently not deserve further investigation as a single agent in this setting.

MiMe, by assessing metabolic response early during the treatment course, will hopefully provide useful information about the drug activity in various cancer types, and about mechanisms of resistance through a potential ambitious translational research program with serial collection of circulating-tumour DNA (ct-DNA).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old
2. Female or male
3. ECOG performance status ≤ 1
4. Life expectancy of greater than 12 weeks
5. Must have histologically confirmed cancer corresponding to the predefined tumour subtypes (esophageal adenocarcinoma, esophageal squamous cell carcinoma, cholangiocarcinoma, urothelial cancer (progressive after immunotherapy), endometrial cancer) and metastatic or non-resectable and refractory to standard platinum regimens (and progressive after immunotherapy for the urothelial cancer).
6. Presence of at least one metabolically measurable tumour lesion on FDG-PET/CT, according to PERCIST. If previously irradiated, must have been more than 2 months before the baseline FDG PET/CT.
7. Measurable disease according to RECIST v 1.1
8. Serum pregnancy test (for subjects of childbearing potential) negative
9. Women of childbearing potential must agree to the use a highly effective method of contraception prior to study entry, during the course of the study and at least 3 months after the last administration of study treatment.
10. Men with childbearing potential partner must agree to use condom during the course of this study and for at least 3 months after the last administration of the study treatment.
11. Adequate coagulation: International Normalized Ratio (INR) ≤ 1.5 x ULN unless subject is receiving anticoagulant therapy as long as INR and activated partial thromboplastin time [aPTT] are within therapeutic range of intended use of anticoagulants
12. Adequate bone marrow function as defined below:

    * Hemoglobin ≥ 10 g/dL
    * Absolute neutrophil count ≥ 1500/µL or 1.5x109/L
    * Platelets ≥ 100000/µL or 100x109/L
    * Leukocytes ≥ 3,000/µL
13. Adequate liver function as defined below:

    * Serum total bilirubin within 1.5 × normal institutional limits (except for Gilbert syndrome where direct bilirubin should be <1.5 institutional ULN)
    * AST/ALT/ALP) levels < 3 × institutional upper limit of normal (or ALT and AST <5 times upper limit of normal if liver metastases are present).
14. Adequate renal function as defined below: Cockcroft-Gault creatine clearance >50ml/min
15. Completion of all necessary screening procedures
16. Ability to swallow capsules
17. Grade ≤ 1 toxicity due to any previous cancer therapy according to the National Cancer Institute Common Terminology Criteria of Adverse Events (NCI-CTCAE, v.4.03). Grade 2 is allowed in case of alopecia and peripheral sensory neuropathy
18. Availability of primary archived tumour tissue block (1 FFPE tumour tissue)
19. Signed Informed Consent form (ICF) obtained prior to any study related procedure

Exclusion Criteria:

1. Subjects meeting one of the following criteria are not eligible for this studyParticipants who have had chemotherapy, radiotherapy, immunotherapy, or targeted therapy within 3 weeks prior study enrolment
2. Participants receiving concomitantly any other experimental agents
3. Patients who have received prior therapy with other CDK4/6 inhibitors
4. Subjects with known brain metastasis; unless the metastasis are asymptomatic and have been stable since at least 2 months prior to treatment start.
5. Patient with meningeal carcinomatosis
6. Have had major surgery within 28 days prior to the start of the treatment to allow for post-operative healing of the surgical wound
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition
8. Bleeding diathesis, thromboembolic event, history of cardiovascular ischemic disease or cerebrovascular incident within the last six months
9. Uncontrolled concurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia
10. Substance abuse, psychiatric illness/social situations, any psychological, familial, sociological, geographical condition, significant medical or surgical condition currently uncontrolled by treatment that would limit compliance with study requirements or interfere with the patient's ability to understand informed consent and participation in the study
11. Pregnant and/or lactating women
12. Uncontrolled Diabetes
13. Known history of HIV infection, or active hepatitis B or C requiring treatment with anti-viral therapy
14. Have received recent (within 28 days prior the enrolment) yellow fever vaccination
15. Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free and are deemed by the investigator to be at low risk for recurrence of that malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Evaluate the anti-tumour activity of abemaciclib in the five tumour types studied in this trial using FDG-PET/CT during the first cycle of therapy (early FDG- PET/CT). | 2 months
  Therapy success rate defined as: PERCIST 15%-assessed Metabolic Response at early FDG-PET/CT (D12-D16)
Evaluate the anti-tumour activity of abemaciclib in the five tumour types studied in this trial using RECISTv1.1 after 2 cycles of therapy as a screening tool. | 2 Months
  Therapy success rate defined as: RECISTv1.1-assessed Disease Control (DC) after 2 treatment cycles (CR or PR or SD)

SECONDARY OUTCOMES:
Evaluate Progression-free survival (PFS define as the time from treatment start until disease progression or death) at 24 weeks from treatment start | 6 months
  RECIST v1.1-based radiological response assessment performed at 24 weeks from the treatment start to determine the PFS
Evaluate Overall Survival (OS defined as the time from treatment start until death) at 24 weeks from treatment start | 6 months
  RECIST v1.1-based radiological response assessment performed at 24 weeks from the treatment start to determine the OS.
To evaluate median progression-free survival (PFS) | 42 months
  Progression Free Survival
Evaluate median overall survival (OS) | 42 months
  Overall Survival
To evaluate toxicity profile | 6 months
  Toxicity profile according to CTCAE version 4.03
Evaluate the correlation of early metabolic response using FDG-PET/CT with morphological response to treatment assessed by RECIST | 6 months
  RECIST v1.1-based radiological response assessment performed at 24 weeks from the treatment start to determine the PFS and OS

CONTACTS AND LOCATIONS:
Overall Officials: Laura Polastro, MD, Study Chair — Jules Bordet Institute
Locations (11):
- Belgium (6):
  - Universitair Ziekenhuis, Antwerp
  - Institut Jules Bordet, Brussels
  - Algemeen Ziekenhuis Groeninge, Kortrijk
  - CHC Saint-Joseph, Liège
  - CHU Ambroise Paré, Mons
  - CHU UCL Namur Sainte-Elisabeth, Namur
- France (5):
  - Centre Oscar Lambret, Lille
  - Institut Paoli-Calmettes, Marseille
  - Centre Henri Becquerel, Rouen
  - Hôpital universitaire de Strasbourg - ICANS, Strasbourg
  - IUCT Oncopole - Institut Claudius Regaud, Toulouse

IPD SHARING:
Plan to Share IPD: No